CLINICAL TRIAL: NCT01459107
Title: Human Upper Extremity Allotransplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00046418
Record Dates: First submitted 2011-09-29; First posted 2011-10-25 (Estimated); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Amputation, Traumatic; Wounds and Injuries; Hand Injuries
Keywords: Hand Transplant; Composite Tissue Allotransplantation (CTA); Vascularized Composite Allotransplantation (VCA); Composite Tissue; Amputation; Upper limb; Immunosuppression
MeSH Terms: conditions — Amputation, Traumatic; Wounds and Injuries; Hand Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Transplantation) (Experimental): Hand/arm transplantation in combination with a novel donor bone marrow cell-based therapy followed by single-drug immunosuppression with potential weaning.
  Interventions: Procedure: Deceased donor hand transplantation; Drug: Bone marrow cell-based therapy & single-drug immunosuppression.

INTERVENTIONS:
Procedure: Deceased donor hand transplantation — Deceased donor hand is surgically attached to recipient arm's stump.
Drug: Bone marrow cell-based therapy & single-drug immunosuppression. — This protocol uses a novel bone marrow cell-based therapy for composite tissue allotransplantation (CTA) rather than conventional triple-drug immunosuppression to facilitate long-term graft survival of deceased donor human upper extremities under low-dose maintenance immunosuppression. Initial T-cell depletion with alemtuzumab is followed by upper extremity transplantation and tacrolimus maintenance therapy. Donor bone marrow cells are infused on Day 10 (±4 days) post-transplantation to elicit a host alloimmune response triggering exhaustion and deletion of the respective host (anti-donor) lymphocyte clones. Subsequently, tacrolimus therapy is given for at least 6 months before spaced weaning is considered in stable recipients.

SUMMARY:
Background: Millions of people each year sustain injuries, have tumors surgically removed, or are born with defects that require complex reconstructive surgeries to repair. In the case of hand, forearm, or arm amputation, prostheses only provide less than optimal motor function and no sensory feedback. However, hand and arm transplantation is a means to restore the appearance, anatomy, and function of a native hand. Although over 70 hand transplants have been performed to date and good functional results have been achieved, widespread clinical use has been limited due to adverse effects of life-long and high-dose immunosuppression needed to prevent graft rejection. Risks include infection, cancer, and metabolic problems, all of which can greatly affect recipients' quality of life, make the procedure riskier, and jeopardize the potential benefits of hand transplantation.

Study Design: This non-randomized, Phase II clinical trial will document the use of a new immunomodulatory protocol (aka - Pittsburgh Protocol, Starzl Protocol) for establishing hand transplantation as a safe and effective reconstructive treatment for upper extremity amputations by minimizing maintenance immunosuppression therapy in unilateral and bilateral hand/forearm transplant patients. This protocol combines lymphocyte depletion with donor bone marrow cell infusion and has enabled graft survival using low doses of a single immunosuppressive drug followed by weaning of treatment. Initially designed for living-related solid organ donation, this regimen has been adapted for use with grafts donated by deceased donors. The investigators propose to perform 30 human hand transplants employing this novel protocol.

Specific Aims: 1) To establish hand transplantation as a safe and effective reconstructive strategy for the treatment of upper extremity amputations; 2) To reduce the risk of rejection and enable allograft survival while minimizing the requirement for long-term high dose multi-drug immunosuppression.

Significance of Research: Hand transplantation could help upper extremity amputees recover functionality, self-esteem, and the capability to reintegrate into family and social life as "whole" individuals. The protocol offers the potential for minimizing the morbidity of maintenance immunosuppression, thereby beneficially shifting the risk/benefit ratio of this life-enhancing procedure and enabling widespread clinical application of hand transplantation.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Recent (≥6 months) or remote (i.e., several decades) unilateral or bilateral upper limb loss (below the shoulder) desiring limb transplantation.
* Below-shoulder amputation.
* Functionless or minimally functional hand desiring removal of functionless / minimally functional hand followed by transplantation.
* Male or female and of any race, color or ethnicity.
* Aged 18-69 years.
* Completes the protocol informed consent form.
* No co-existing medical condition which, in the opinion of the study team, could affect the immunomodulatory protocol, surgical procedure, or functional results (see Donor and Recipient Exclusion Criteria below. If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of upper extremity transplantation.)
* No co-existing psycho-social problems (i.e., alcoholism, drug abuse).
* Negative for malignancy for past 5 years.
* Negative for HIV at transplant.
* Negative crossmatch with donor.
* If female of child-bearing potential, negative serum pregnancy test.
* If female of child-bearing potential, consent to use reliable contraception for at least one year following transplantation.
* Consents to bone marrow infusion as part of the treatment regime.
* USA citizen or equivalent, or foreigner with documentation of ability to pay for transplant and required follow-up care.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regime.

Donor Inclusion Criteria:

Donors will be selected by the upper extremity transplant team in conjunction with the organ procurement organization (OPO) according to the following criteria:

* Brain dead meeting the criteria for Determination of Death.
* Family consent for limb donation.
* Stable donor (i.e., does not require excessive vasopressors to maintain blood pressure).
* Aged 16 - 65 years.
* Limb matched for size with recipient.
* Same blood type as recipient.
* Negative lymphocytotoxic crossmatch.
* Accurately matched for gender, skin tone, and race (relative requirements depending on recipient consent).

Exclusion Criteria:

• Positive for any of the following conditions:

* Untreated sepsis.
* HIV (active or seropositive).
* Active tuberculosis.
* Hepatitis B or C.
* Viral encephalitis.
* Toxoplasmosis.
* Malignancy (within past 5 years).
* Current/recent (within 3 months of donation/screening consent) IV drug abuse.
* Paralysis of ischemic or traumatic origin.
* Inherited peripheral neuropathy.
* Infectious, post infectious, or inflammatory (axonal or demyelinating) neuropathy.
* Toxic neuropathy (i.e. heavy metal poisoning, drug toxicity, industrial agent exposure).
* Mixed connective tissue disease.
* Severe deforming rheumatoid or osteoarthritis in the limb.

Donor Only:

• Tattoos:

* Non-professional tattoo within last 6 months, or
* Personally identifiable tattoo (i.e., donor name) on potential transplant.

Recipient Only:

* Type I (insulin-dependent) diabetes mellitus
* Conditions that, in the opinion of the study team, may impact the immunomodulatory protocol potentially exposing the recipient to an unacceptable risk under immunosuppressive treatment.
* Sensitized recipients with high levels (50%) of panel-reactive human leukocyte antigen (HLA) antibodies.
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Mixed connective tissue diseases and collagen diseases can result in poor wound healing after surgery.
* Conditions that may impact functional outcomes including Lipopolysaccharidosis and amyloidosis (may impact nerve regeneration) or rare disorders of bone healing like osteopetrosis.
* Patients considered unsuitable per the consulted Psychiatrists appraisal.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07-21 (Actual); Primary Completion 2036-06-30 (Estimated); Study Completion 2036-06-30 (Estimated)

PRIMARY OUTCOMES:
Graft Survival | Transplantation through end of study period (up to 5 years)
  Post-operative graft survival will be documented monthly Months 1-12 and quarterly (every 3 months) Years 2-5.

SECONDARY OUTCOMES:
Documentation of immunosuppression required by transplanted participants to maintain graft. | Transplantation to end of study period (up to 5 years)
  Post-operative serum trough levels will be documented daily Days 1-28, semiweekly Weeks 5-12, weekly Weeks 13-25, biweekly Weeks 26-38, monthly Months 10-12, and quarterly (every 3 months) Years 2-5.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Cooney, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Pooled patient data will be shared.

REFERENCES:
- [Background] Schneeberger S, Gorantla VS, Brandacher G, Zeevi A, Demetris AJ, Lunz JG, Metes DM, Donnenberg AD, Shores JT, Dimartini AF, Kiss JE, Imbriglia JE, Azari K, Goitz RJ, Manders EK, Nguyen VT, Cooney DS, Wachtman GS, Keith JD, Fletcher DR, Macedo C, Planinsic R, Losee JE, Shapiro R, Starzl TE, Lee WP. Upper-extremity transplantation using a cell-based protocol to minimize immunosuppression. Ann Surg. 2013 Feb;257(2):345-51. doi: 10.1097/SLA.0b013e31826d90bb. PMID 23001085
- See also: Study website including additional related information. — https://www.hopkinsmedicine.org/transplant/programs/reconstructive-transplant/hand-arm-transplant